CLINICAL TRIAL: NCT03744923
Title: Perioperative Analgesia for Flank Incision Surgeries
Brief Title: Quadratus Lumborum Block (Transmuscular Approach) VS. TransversusAbdominus Plane Block(Unilateral Posterior Approach) for Perioperative Analgesia in Patients Undergoing Flank Incision Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, principal investigator, Cairo University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: N-36-2018
Record Dates: First submitted 2018-11-08; First posted 2018-11-19 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transmuscular QLB group (Active Comparator): Ultrasound device will be used; The probe is placed in the mid-axillary line cranially to the iliac crest to identify the three muscles of the anterior abdominal wall Then, scan dorsally keeping the transverse orientation until observing that the transverse abdominus muscle becomes aponeurotic, and this aponeurosis is followed until the QL muscle is clearly visualized with its attachment to the lateral edge of the transverse process of the L2 vertebral body and visualize the thoracolumbar fascia The needle (20G spinal needle) is inserted in-plane from posterior to anterior and the tip of the needle is advanced towards then through the QL muscle, penetrating the ventral proper fascia of the QL muscle. The target site for injection is the plane between quadratus lumborum and psoas major. This will be followed by injection of Bupivacaine 0.5 % (0.25ml/kg) and lidocaine 2% (0.15ml/kg) mixed together.
  Interventions: Procedure: transmuscular QL block
- unilateral posterior TAP block group (Active Comparator): under ultrasonographic guidance,the probe will be positioned transversely midway between the iliac crest and the costal margin at level of mid axillary line.
  Once the external oblique muscle (EOM), internal oblique muscle (IOM) and transversus abdominis muscle (TAM) are visualized at the level of the mid-axillary line between the 12th rib and the iliac crest, the puncture area and the ultrasound probe were prepared in a sterile manner. After identification of the neuro-facial plane between IOM and TAM, the block was performed with the 20G spinal needle. The needle will be directed to approach the TAP with "in-plane" USG-guided technique. Once the tip of the needle placed in the space between the IOM and TAM, Inject a 1 ml test dose of lidocaine 2% for hydro visualization of needle-tip position and confirming its correct positioning. This will be followed by injection of Bupivacaine 0.5 % (0.25ml/kg) and lidocaine 2% (0.15ml/kg) mixed together.
  Interventions: Procedure: Transversus Abdominus Plane block
- control group (No Intervention): the patients will not receive any blocks

INTERVENTIONS:
Procedure: transmuscular QL block — Ultrasound device will be used; The probe is placed in the mid-axillary line cranially to the iliac crest to identify the three muscles of the anterior abdominal wall. Then, scan dorsally keeping the transverse orientation until observing that the transversusabdominus muscle becomes aponeurotic, and this aponeurosis is followed until the QL muscle is clearly visualized with its attachment to the lateral edge of the transverse process of the L2 vertebral body and visualize the thoracolumbar fascia at the lateral edge of the QL muscle.
  The view of the psoas major muscle (PM) anteriorly, the erector spinae muscle (ESM) posteriorly and the QL muscle adherent to the apex of the transverse process result in a well recognizable pattern of a Shamrock with three leaves (trifoliate).
  Arms: Transmuscular QLB group
Procedure: Transversus Abdominus Plane block — Posterior TAP block will be performed on the same side of surgery (unilateral) under ultrasonographic guidance with a with broadband (7-13MHz) linear probe covered with a sterile plastic sheath. Probe will positioned transversely midway between the iliac crest and the costal margin at level of mid axillary line.
  Once the external oblique muscle (EOM), internal oblique muscle (IOM) and transversus abdominis muscle (TAM) are visualized at the level of the mid axillary line between the 12th rib and the iliac crest, the puncture area and the ultrasound probe were prepared in a sterile manner. After identification of the neuro-facial plane between IOM and TAM, block was performed with 20G spinal needle. The needle will be directed to approach the TAP with "in-plane" USG-guided technique. Once the tip of the needle placed in the space between the IOM and TAM, Inject a 1 ml test dose of lidocaine 2% for hydrovisualization of needle-tip position and confirming its correct postioning.
  Arms: unilateral posterior TAP block group

SUMMARY:
Severe perioperative pain experienced after surgical procedures performed by flank incision is mainly related to incision of many muscles. Postoperative pain affects patient comfort, satisfaction, prolongs the duration of hospital stay and increases post-procedure complications. This study is designed to compare the success rate of Unilateral Ultrasound Guided Transmuscular Quadratus Lumborum Block with Unilateral posterior Ultrasound Guided TransversusAbdominus Plane block in providing perioperative analgesia in Patients undergoing Flank Incision surgeries in the Urosurgery Theater at KasrAlainy University Hospitals.

DETAILED DESCRIPTION:
Patients aged from 20-60 years old, scheduled for flank surgery procedure will be included in the study. Patients will be randomly allocated using concealed closed envelope method into one of three groups:

Group A (n=16): will receive USG TransmuscularQLB after induction of general anesthesia.

Group B (n=16): will receive unilateral USG posterior TAP Block after induction of General anesthesia.

Group C (n=16): (control group) will not receive any blocks.general anesthesia will be induced using propofol 2-3 mg/kg over 20-30 seconds, fentanyl 2 µg/kg, and atracurium 0.5 mg/kg to facilitate endotracheal intubation. Anesthesia will be maintained using isoflurane 1.5 %, atracurium at a dose of 0.1 mg/kg every 20 minutes. For all patients, fluid management will be strict according to body weight and blood loss will be adequately estimated and replaced. In the three groups, the observing anesthetist will be advised to give fentanyl increment doses (0.5 µg/kg) when mean blood pressure, heart rate or both increased by more than 20% from the baseline, lacrimation or sweating (signs of inadequate analgesia).

Postoperatively, all patients will receive IV paracetamol 1gm every 8 hours. As a rescue analgesic, meperidine (0.5 mg/kg) will be used when VAS score > 4. The following data will be recorded1- Duration of the surgery 2- Time required to perform the blocks in minutes 3- Intraoperative mean blood pressure and heart rate will be recorded in all groups immediately after induction, at the surgical incision and every 15 minutes till the end of the procedure.

4- Total amount of intraoperative fentanyl consumption will be recorded 5- Immediate postoperative blood pressure and heart rate will be recorded 6- Visual Analogue scale (VAS) for pain will be applied postoperatively at rest and during movement. Pain will be assessed with a 10-cm ruler ranging from no pain (0) to severe pain (10). Evaluation will be performed immediately postoperative, at 30 minutes, 1 hour, 2 hours, 4 hours, 6hours and 12 hours postoperatively.

7- The time of the first analgesic request (rescue analgesia) in the postoperative period will be recorded (defined as the time between the end of surgery and the request of the first dose of postoperative analgesics). As a rescue analgesic, meperidine (0.5 mg/kg) will be used when VAS score > 4.

8- Postoperative nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

* Patients age between >20 and <60.
* Patients scheduled for Urological flank surgery (open nephrectomy)
* Ability to sign the consent
* ASA classification I, II
* Body Mass Index (BMI) < or = 30
* Duration of surgery less than 3 hours

Exclusion Criteria:

* Refusal of the regional block.
* Bleeding disorders (INR >1.4 )( platelet count <100,000/mm3 )
* Skin lesions or infection at the site of proposed needle insertion.
* Evidence of peritonitis or septicemia.
* Hepatic disease e.g. liver cell failure or hepatic malignancy or hepatic enlargement.
* Patients with ventriculoperitoneal shunts in situ.
* Allergy to amide local anesthetics, fentanyl or meperidine.
* Patients suffering from neurological disease.
* ASA classification > II
* BMI > 30
* Duration of surgery more than 3 hours

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
fentanyl consumption in the intraopertive period | 3 hours
  Measurement of total the amount of fentanyl consumption in the intraopertive period in the three allocated groups as indicator for hemodynamic stability and efficacy of both types of blocks.

SECONDARY OUTCOMES:
doses of postoperative mepridine analgesics | 24 hours
  as an indication of success of the blocks postoperatively
VAS(visual analogue score) | 24 hours
  visual analogue scale for pain assessment postopertively Pain will be assessed with a 10-cm ruler ranging from no pain (0) to severe pain (10).

CONTACTS AND LOCATIONS:
Overall Officials: kasr alaini hospital, Study Director — Cairo University
Locations (1):
- Amany Hassan Saleh, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saleh AH, Abdallah MW, Mahrous AM, Ali NA. Quadratus lumborum block (transmuscular approach) versus transversus abdominis plane block (unilateral subcostal approach) for perioperative analgesia in patients undergoing open nephrectomy: a randomized, double-blinded, controlled trial. Braz J Anesthesiol. 2021 Jul-Aug;71(4):367-375. doi: 10.1016/j.bjane.2021.01.009. Epub 2021 Mar 21. PMID 33762197